CLINICAL TRIAL: NCT00760435
Title: Infliximab (Remicade®) Plus Intravenous Immunoglobulin (IVIG) for the Primary Treatment of Patients With Acute Kawasaki Disease
Brief Title: Infliximab Plus Intravenous Immunoglobulin for the Primary Treatment of Kawasaki Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Jane C. Burns, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01FD003514-01 (FDA)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; Infliximab; Remicade; Pediatrics
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Infliximab plus Intravenous immunoglobulin (IVIG)
  Interventions: Drug: Infliximab
- 2 (Placebo Comparator): Placebo plus IVIG
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — 5 mg/kg IV over 2 hours once
  Other Names: Remicade
  Arms: 1
Drug: Placebo — Placebo (same volume as active drug)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the addition of infliximab to standard primary therapy of intravenous immunoglobulin (IVIG) and high dose aspirin will reduce resistance to therapy in acute Kawasaki disease (KD).

DETAILED DESCRIPTION:
KD, an orphan disease of low prevalence in U.S. children, causes significant long term cardiac sequelae in a subset of patients. KD patients that are resistant to therapy are more likely to develop coronary artery abnormalities. This phase III placebo-controlled, multicenter, randomized clinical trial of infliximab plus standard therapy vs. placebo plus standard therapy in acute KD will determine if the addition of infliximab to primary therapy can reduce the percentage of children resistant to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. All eligible subjects, or legal representative, must provide written informed consent/assent, prior to initiation of any study procedure.
2. Eligible subjects will be infants and children, 4 weeks to 17 years old, who have had fever for 3 to 15 days (illness day 1 = first day of fever ≥ 38.3° C)
3. Patients who meet one of the following sets of criteria will be eligible for enrollment (adapted from AHA guidelines: Newburger et al. 2004):

   * Case definition for complete KD: Fever (≥ 38.3°C) for ≥ 3 days and 4/5 standard clinical criteria (Table 1)
   * Case definition for incomplete KD: Fever ≥ 5 days and 2-3 clinical criteria plus either C-reactive protein (CRP) ≥ 3.0 mg/dL or ESR ≥40 mm/hr AND ≥ 3 supplemental laboratory criteria: albumin ≤ 3.0 g/dl, anemia for age, ALT ≥ 45, platelet count ≥ 450,000/mm3, white blood cell count ≥ 15,000/mm3, or urinalysis with ≥10 white blood cells/hpf.
   * Case definition for incomplete KD with echocardiogram data: Fever ≥ 5 days and <4/5 clinical criteria plus abnormal echocardiogram with z score of LAD or RCA ≥ 2.5
4. Females of childbearing potential and males must be using adequate contraception (abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) throughout the trial.
5. All eligible subjects must have a chest radiograph within one week prior to first infusion of study drug with no evidence of tuberculosis or other infection.

Exclusion Criteria:

1. Have been receiving corticosteroids (i.e. via any route) at doses > 1 mg/kg prednisone equivalent daily.
2. History of tuberculosis (TB) or TB exposure.
3. Have received a BCG vaccination within the past 6 months.
4. History of histoplasmosis or coccidioidomycosis
5. Have received anakinra (Kineret®), etanercept (Enbrel®), or adalimumab (Humira®) within 1 month prior to first study drug administration.
6. Have any chronic disease, except asthma, atopic dermatitis or controlled seizure disorder.
7. Have documented history of current active Hepatitis B or a history of Hepatitis C infection.
8. Have a documented history of human immunodeficiency virus (HIV) infection.
9. Have received a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to the first study drug administration).
10. Have a known malignancy or history of malignancy within the 5-year period prior to first study drug administration (with the exception of basal cell or squamous cell carcinoma of the skin that has been completely excised without evidence of recurrence).
11. Have a history of prior lymphoproliferative disease including lymphoma.
12. Have multiple sclerosis or other central demyelinating disorder.
13. Have received any previous treatment with infliximab or other monoclonal antibodies
14. Have used any investigational drug within 1 month prior to first study drug administration or within 5 half-lives of the investigational agent, whichever is longer.
15. Are participating in another investigative trial, involving investigational agents, during participation in this trial.
16. Have a history of substance abuse (drug or alcohol) within the previous 3 years.
17. Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.
18. Have a known allergy to murine proteins or other chimeric proteins.
19. Patients with ischemic congestive heart failure, defined by ECG changes, elevated Troponin 1 and CPK-MB consistent with myocardial ischemia.
20. Have an abnormal chest radiograph
21. Afebrile for ≥ 48 hours

Ages: 4 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Burns, M.D., Principal Investigator — University of California, San Diego; Adriana H. Tremoulet, M.D., Study Director — University of California, San Diego; Octavio Ramilo, M.D., Study Director — University of Texas
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Background] Burns JC, Best BM, Mejias A, Mahony L, Fixler DE, Jafri HS, Melish ME, Jackson MA, Asmar BI, Lang DJ, Connor JD, Capparelli EV, Keen ML, Mamun K, Keenan GF, Ramilo O. Infliximab treatment of intravenous immunoglobulin-resistant Kawasaki disease. J Pediatr. 2008 Dec;153(6):833-8. doi: 10.1016/j.jpeds.2008.06.011. Epub 2008 Jul 30. PMID 18672254
- [Background] Tremoulet AH, Best BM, Song S, Wang S, Corinaldesi E, Eichenfield JR, Martin DD, Newburger JW, Burns JC. Resistance to intravenous immunoglobulin in children with Kawasaki disease. J Pediatr. 2008 Jul;153(1):117-21. doi: 10.1016/j.jpeds.2007.12.021. Epub 2008 Mar 4. PMID 18571548
- [Background] Newburger JW, Sleeper LA, McCrindle BW, Minich LL, Gersony W, Vetter VL, Atz AM, Li JS, Takahashi M, Baker AL, Colan SD, Mitchell PD, Klein GL, Sundel RP; Pediatric Heart Network Investigators. Randomized trial of pulsed corticosteroid therapy for primary treatment of Kawasaki disease. N Engl J Med. 2007 Feb 15;356(7):663-75. doi: 10.1056/NEJMoa061235. PMID 17301297
- [Background] Newburger JW, Takahashi M, Gerber MA, Gewitz MH, Tani LY, Burns JC, Shulman ST, Bolger AF, Ferrieri P, Baltimore RS, Wilson WR, Baddour LM, Levison ME, Pallasch TJ, Falace DA, Taubert KA; Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease, Council on Cardiovascular Disease in the Young, American Heart Association. Diagnosis, treatment, and long-term management of Kawasaki disease: a statement for health professionals from the Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease, Council on Cardiovascular Disease in the Young, American Heart Association. Pediatrics. 2004 Dec;114(6):1708-33. doi: 10.1542/peds.2004-2182. PMID 15574639
- [Background] Burns JC, Mason WH, Hauger SB, Janai H, Bastian JF, Wohrley JD, Balfour I, Shen CA, Michel ED, Shulman ST, Melish ME. Infliximab treatment for refractory Kawasaki syndrome. J Pediatr. 2005 May;146(5):662-7. doi: 10.1016/j.jpeds.2004.12.022. PMID 15870671
- [Derived] Tremoulet AH, Jain S, Jaggi P, Jimenez-Fernandez S, Pancheri JM, Sun X, Kanegaye JT, Kovalchin JP, Printz BF, Ramilo O, Burns JC. Infliximab for intensification of primary therapy for Kawasaki disease: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet. 2014 May 17;383(9930):1731-8. doi: 10.1016/S0140-6736(13)62298-9. Epub 2014 Feb 24. PMID 24572997
- [Derived] Burns JC, Song Y, Bujold M, Shimizu C, Kanegaye JT, Tremoulet AH, Franco A. Immune-monitoring in Kawasaki disease patients treated with infliximab and intravenous immunoglobulin. Clin Exp Immunol. 2013 Dec;174(3):337-44. doi: 10.1111/cei.12182. PMID 23901839
- [Derived] Kanegaye JT, Van Cott E, Tremoulet AH, Salgado A, Shimizu C, Kruk P, Hauschildt J, Sun X, Jain S, Burns JC. Lymph-node-first presentation of Kawasaki disease compared with bacterial cervical adenitis and typical Kawasaki disease. J Pediatr. 2013 Jun;162(6):1259-63, 1263.e1-2. doi: 10.1016/j.jpeds.2012.11.064. Epub 2013 Jan 7. PMID 23305955

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab Arm: 98 recieved infliximab plus IVIG
  Infliximab: 5 mg/kg IV over 2 hours once
- Placebo Arm: 98 received Placebo plus IVIG
  Placebo: Placebo (same volume as active drug)
Period: Overall Study
Arm/Group | Infliximab Arm | Placebo Arm
Started | 98 | 98
Completed | 94 | 93
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab Arm | Placebo Arm | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.0 [1.9 to 4.8] | 2.8 [1.8 to 4.2] | 2.9 [1.8 to 4.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 60 | 61 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 14 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 8 | 18
  White | 61 | 59 | 120
  More than one race | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 64 | 121
  Not Hispanic or Latino | 41 | 34 | 75
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 98 | 98 | 196

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects in Each Arm That Have Persistent or Recrudescent Fever 24 Hours After Completion of the Intravenous Immunoglobulin (IVIG) Infusion
Time Frame: 10 weeks
Population: 1 subject in the placebo group was removed from the modified ITT analysis (this subject was removed from the study prior to receiving the placebo)
Measure: Number; unit: participants
Groups:
- Infliximab: 98 subjects treated with infliximab + IVIG
- Placebo: 97 subjects who received placebo + IVIG
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 98 | 97
participants | 11 | 11

2. Secondary Outcome: Number of Days of Fever Following Therapy During Study Period (up to 6 Weeks)
Time Frame: up to 6 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 98 | 97
days | 1 [1 to 2] | 2 [1 to 2]

3. Secondary Outcome: Change in C-reactive Protein (CRP) From Baseline at 24 Hours After Completion of Intravenous Immunoglobulin (IVIG) by Study Arm.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 98 | 97
mg/dL | -6.6 [-7.7 to -5.4] | -3.6 [-4.8 to -2.5]

4. Secondary Outcome: Change From Baseline in Left Anterior Descending Coronary Artery Outcomes at Week 2 by Treatment Arm
Description: left anterior descending coronary artery Z-score; a Z score is the coronary artery adjusted for body surface area
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 98 | 97
Z-score | -0.605 [-0.808 to -0.403] | -0.313 [-0.514 to -0.111]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Infliximab Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 22/98 | 17/98
Other Adverse Events (participants affected / at risk) | 49/98 | 61/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Infliximab Arm (N=98) | Placebo Arm (N=98)
Fever (Immune system disorders) | 11 (11) | 11/97 (11) — Fever
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Coronary artery abnormality (Cardiac disorders) | 6 (6) | 2 (2) — CAA that warranted prolonged hospitalization
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Macrophage Activation Syndrome (Immune system disorders) | 0 (0) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
URI (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab Arm (N=98) | Placebo Arm (N=98)
IVIG Infusion Reaction (Immune system disorders) | 0 (0) | 13 (13) — Hypotension or chills during IVIG infusion
Coronary artery abnormality (Cardiac disorders) | 5 (5) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10)
URI (Infections and infestations) | 16 (16) | 19 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Vomiting/nausea/abdominal pain (Gastrointestinal disorders) | 9 (9) | 17 (17)
Worsening of WBC (Blood and lymphatic system disorders) | 10 (10) | 13 (13)

LIMITATIONS AND CAVEATS:
The major limitation of our study was the low rate of treatment-resistance in the placebo arm (11%, compared to historical IVIG resistance rates of 20%), which decreased our power to detect a difference in the primary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No